CLINICAL TRIAL: NCT01874132
Title: A Randomised Longitudinal Study of Exercise Prescription for Older Adults: Mode and Intensity to Induce the Highest Cardiovascular Health-related Benefits
Brief Title: Study of the Long-term Effects of Exercise on Heath Indicators in Older People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Trás-os-Montes and Alto Douro (Other)
Responsible Party: Principal Investigator, Nelson Joaquim Fortuna de Sousa, Professor, University of Trás-os-Montes and Alto Douro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CVD-2009-EX
Record Dates: First submitted 2013-06-06; First posted 2013-06-10 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-03

CONDITIONS: Hypertension With Complications and Secondary Hypertension; Overweight and Obesity; Lipid Metabolism Disorders; Sarcopenia; Osteoporosis; Personal Satisfaction
Keywords: Exercise; Blood pressure; Lipids; Body composition; Fitness; Bone density; Quality of life
MeSH Terms: conditions — Overweight; Obesity; Lipid Metabolism Disorders; Sarcopenia; Osteoporosis; Personal Satisfaction; Motor Activity | interventions — Exercise; Resistance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Aerobic exercise training (Experimental): Dose response
  Interventions: Behavioral: Exercise training
- Aerobic and resistance exercise training (Experimental): Dose response
  Interventions: Behavioral: Exercise training
- Control (No Intervention): Non-exercising control group

INTERVENTIONS:
Behavioral: Exercise training — Both training programs were of moderate-to-vigorous intensity, three days per week for nine months.
  Other Names: Aerobic training; resistance training; Combined training; multicomponent training
  Arms: Aerobic and resistance exercise training; Aerobic exercise training

SUMMARY:
Cardiovascular diseases (CVD) represent the most frequent cause of death among the elderly population. Hypertension, unfavorable lipid profile, obesity and physical inactivity are among the main risk factors for CVD. In contrast, mortality from CVD is inversely related to levels of physical activity, and is lower in individuals who exercise and have higher functional fitness levels. Thus, the Centers for Disease Control and Prevention, the American College of Sports Medicine, and the American Heart Association have recommended 20-30 min of moderate-to-vigorous aerobic training for the elderly, preferably every day or at least 3 days a week in the case of vigorous exercise.The same organizations also suggest the inclusion of resistance training in order to improve functional fitness. Therefore, the purpose of this study was to compare different exercise modalities in long-term changes of CVD risk factors and physical fitness among older adults.

ELIGIBILITY:
Inclusion Criteria:

* Older adults living independently;
* medical approval.

Exclusion Criteria:

* Non-smokers;
* Non-morbidly obese;
* No history of severe hypertension;
* No history of falls;
* No orthopaedic, neurological, pulmonary, or cardiac problems.

Ages: 65 Years to 79 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 66 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Sousa, PhD, Principal Investigator — Research Center in Sport Sciences, Health Sciences and Human Development; University of Trás-os-Montes e Alto Douro; José Oliveira, PhD, Study Director — Research Center in Physical Activity, Health and Leisure; Sport Faculty, University of Porto; Romeu Mendes, MD, Study Chair — University of Trás-os-Montes and Alto Douro
Locations (1):
- Maia City Council facilities, Maia, Portugal

REFERENCES:
- [Background] Sousa N, Mendes R, Oliveira J. Response to Drs. Safer and Safer. J Am Geriatr Soc. 2014 Mar;62(3):590-1. doi: 10.1111/jgs.12712. No abstract available. PMID 24628645
- [Result] Sousa N, Mendes R, Abrantes C, Sampaio J, Oliveira J. Long-term effects of aerobic training versus combined aerobic and resistance training in modifying cardiovascular disease risk factors in healthy elderly men. Geriatr Gerontol Int. 2013 Oct;13(4):928-35. doi: 10.1111/ggi.12033. Epub 2013 Feb 26. PMID 23441809
- [Result] Sousa N, Mendes R, Abrantes C, Sampaio J, Oliveira J. A randomized 9-month study of blood pressure and body fat responses to aerobic training versus combined aerobic and resistance training in older men. Exp Gerontol. 2013 Aug;48(8):727-33. doi: 10.1016/j.exger.2013.04.008. Epub 2013 Apr 26. PMID 23628502
- [Result] Sousa N, Mendes R, Abrantes C, Sampaio J, Oliveira J. Is once-weekly resistance training enough to prevent sarcopenia? J Am Geriatr Soc. 2013 Aug;61(8):1423-4. doi: 10.1111/jgs.12387. No abstract available. PMID 23937497
- [Result] Sousa N, Mendes R, Abrantes C, Sampaio J, Oliveira J. Effectiveness of combined exercise training to improve functional fitness in older adults: A randomized controlled trial. Geriatr Gerontol Int. 2014 Oct;14(4):892-8. doi: 10.1111/ggi.12188. Epub 2014 Apr 30. PMID 24779956
- [Result] Sousa N, Mendes R, Abrantes C, Sampaio J, Oliveira J. A randomized study on lipids response to different exercise programs in overweight older men. Int J Sports Med. 2014 Dec;35(13):1106-11. doi: 10.1055/s-0034-1374639. Epub 2014 Jul 10. PMID 25009971
- [Result] Sousa N, Mendes R, Silva A, Oliveira J. Combined exercise is more effective than aerobic exercise in the improvement of fall risk factors: a randomized controlled trial in community-dwelling older men. Clin Rehabil. 2017 Apr;31(4):478-486. doi: 10.1177/0269215516655857. Epub 2016 Jul 10. PMID 27353246

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aerobic Exercise Training | Aerobic and Resistance Exercise Training | Control
Started | 22 | 22 | 22
Completed | 18 | 18 | 19
Not Completed | 4 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aerobic Exercise Training | Aerobic and Resistance Exercise Training | Control | Total
Number analyzed (Participants) | 22 | 22 | 22 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 22 | 22 | 22 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.0 (4.9) | 71.3 (4.6) | 67.2 (5.5) | 69.5 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 22 | 22 | 22 | 66
Region of Enrollment [Number; unit: participants]
  Portugal | 22 | 22 | 22 | 66

OUTCOME MEASURES:

1. Primary Outcome: Cardiovascular Disease Risk Factors
Description: Descriptive frequency of the number of cardiovascular risk factors aggregated in each participant. The risk factors considered were: (i) hypertension; (ii) obesity; and (iii) dyslipidemia.
Time Frame: one year
Population: Only 48 participants completed the body composition, blood pressure and hematology assessments, and were included in analysis.
Measure: Number; unit: participants
Arm/Group | Aerobic Exercise Training | Aerobic and Resistance Exercise Training | Control
Number analyzed (Participants) | 15 | 16 | 17
participants
  0 risk-factors | 3 | 4 | 5
  1 risk-factor | 7 | 5 | 8
  2 risk-factors | 5 | 7 | 4

2. Secondary Outcome: Risk of Falls
Description: Descriptive frequency of the number of participants who took ≥12 seconds to complete the Timed Get-up and Go test, and those who took less than 12 seconds (low risk of falling).
Time Frame: One year
Measure: Count of Participants; unit: Participants
Arm/Group | Aerobic Exercise Training | Aerobic and Resistance Exercise Training | Control
Number analyzed (Participants) | 22 | 22 | 22
Participants
  High risk of fall (TUG≥12 seconds) | 7 | 6 | 5
  Low risk of fall | 15 | 16 | 17

3. Other Pre Specified Outcome: Quality of Life
Description: Measured by the Satisfaction With Life Scale.
Time Frame: One year
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Aerobic Exercise Training | Aerobic and Resistance Exercise Training | Control
Serious Adverse Events (participants affected / at risk) | 1/22 | 2/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aerobic Exercise Training (N=22) | Aerobic and Resistance Exercise Training (N=22) | Control (N=22)
Postural orthostatic hypotension during the study (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Fall during the study (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No